CLINICAL TRIAL: NCT06864637
Title: Nutrition for Trauma (N4T) Community Survey
Brief Title: Nutrition for Trauma Community Survey
Acronym: N4T
Status: Enrolling by invitation | Type: Observational
Sponsor: True Paleo Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 20241101
Record Dates: First submitted 2025-02-27; First posted 2025-03-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Psychological Trauma, Historical; Nutrition; PTSD - Post Traumatic Stress Disorder
Keywords: Psychological Trauma; Nutrition; body-mind-spirit; PTSD - Post Traumatic Stress Disorder; survey
MeSH Terms: conditions — Historical Trauma; Combat Disorders; Psychological Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single group: This is a cross-sectional survey involving a single group of 30-300 participants. The survey aims to gather data on [if participants view and respond to trauma from a holistic perspective through body (nutrition), mind (mental health rejuvenation and renewal), and spirit (faith-based) lens]. There are no distinct groups or follow-up periods.

SUMMARY:
The survey will help investigators learn everything about how people view and respond to trauma from a holistic perspective through body (nutrition), mind (mental health rejuvenation and renewal), and spirit (faith-based) lens. Researchers aim to evaluate if such practices will be effective in helping participants with significant life challenges due to trauma, negative life events, or extremely stressful events will recover from these types of lifestyles. The responses will be used to shape the integrative protocols that the investigators develop for professionals involved with trauma clients. This can help increase recovery rates and lead to productive lives.

DETAILED DESCRIPTION:
What is the purpose of this study?

The study is being done to answer the following question:

Can lack of body-mind-spirit practices heighten psychological trauma and is lack of these practices increased in this population?

The survey will help the investigators learn everything about how people view and respond to trauma from a holistic perspective through body (nutrition), mind (mental health rejuvenation and renewal), and spirit (faith-based) lens. Researchers aim to evaluate if such practices will be effective in helping participants with significant life challenges due to trauma, negative life events, or extremely stressful events will recover from these types of lifestyles. The responses will be used to shape the integrative protocols that the investigators develop for professionals involved with trauma clients. This can help increase recovery rates and lead to productive lives.

What is required? This survey will ask questions related to demographics, past traumatic events, levels of stress, dietary habits, self-care practices, and beliefs surrounding holistic wellness.

ELIGIBILITY:
Inclusion Criteria:

* Any one not listed in exclusion criteria that is over 18 years of age

Exclusion Criteria:

* Must not be a prisoner
* Must not be pregnant
* Must not be under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ‬ Any one not listed in exclusion criteria that is over 18 years of age.
  Participants will fill out surveys at various community locations or online. More in depth-explanation is outlined on the informed‬ consent form. The investigators will not be utilizing this survey in a prison, therefore, prisoners will not be present. The investigators will determine if‬‭ vulnerable populations are present by asking for a government ID to check date of birth and asking a pre-screening question "is the parrticipant currently pregnant?" The informed consent form indicates during the signing process that only adults 18 and older may‬‭ participate.‬
  ‭
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Trauma that Lack of BMS Practices | through study completion, an average of 1 year
  The investigators hypothesize that there will be a strong positive correlation between lack of body-mind-spirit practices and trauma that lead to‬‭ significant life challenges, evidencing the need for community programs tailored to support participants lifestyle‬‭ recovery.‬

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jasmine B Hollywood, DCN, MS, BA-Psy, Principal Investigator — True Paleo Inc.
Locations (1):
- Online, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. This decision is based on privacy and confidentiality concerns to protect the personal information of participants.